CLINICAL TRIAL: NCT06551961
Title: A Randomised Placebo Controlled Trial of Chronic Feeding of INuliN And Methylcellulose On Colonic fermentatioN
Brief Title: Effect of Chronic Feeding of Inulin And Methylcellulose on Colonic Fermentation
Acronym: CINNAMON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: FMHS-199-0524
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: inulin; fermentation; colon; gas
MeSH Terms: conditions — Irritable Bowel Syndrome; Mucopolysaccharidosis IV | interventions — Methylcellulose; Inulin; maltodextrin

STUDY DESIGN:
Intervention Model Description: 2 treatment two period cross-over trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Servings provided in identical pots whose content is only known by one assistant who is not involved in collecting outcomes or analysis of results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- methylcellulose (Active Comparator): 2.5 g of Inulin and 2.5g methylcellulose in 62.5 mL water given thrice daily for 7 days increasing to 5 g of Inulin and 5g methylcellulose in 125 mL water on day 8 continuing until day 14
  Interventions: Dietary Supplement: methylcellulose; Dietary Supplement: inulin
- Placebo (Placebo Comparator): 2.5 g of Inulin and 2.5g maltodextrin in 62.5 mL water given thrice daily for 7 days increasing to 5 g of Inulin and 5g maltodextrin in 125 mL water on day 8 continuing until day 14
  Interventions: Dietary Supplement: inulin; Dietary Supplement: maltodextrin

INTERVENTIONS:
Dietary Supplement: methylcellulose — 2.5 and 5 gm Methylcelllose heated to create a gel
  Other Names: Benecel
  Arms: methylcellulose
Dietary Supplement: inulin — 2.5 and 5 gm inulin powder dissolved in water
Dietary Supplement: maltodextrin — 2.5 and 5gm maltodextrin dissolved in water
  Other Names: Glusidex
  Arms: Placebo

SUMMARY:
To determine the effect on tolerance and gas production from chronic feeding of fermentable fibre (inulin) incorporated into a gel forming fibre (methylcellulose) compared with placebo (maltodextrin)

DETAILED DESCRIPTION:
Our challenge is to understand how various dietary fibres interact to alter colonic fermentation of FODMAPs (fermentable oligosaccharides, disaccharides, monosaccharides and polyols) with the aim of reducing gaseous distension of the colon and hence symptoms. Our previous studies have shown how psyllium, a gel forming natural fibre can reduce gas production induced by a dietary FODMAP inulin when it reaches the colon. The investigators are exploiting a range of food grade modified celluloses which can form gels at body temperature to perform human studies to explore whether the beneficial effect of psyllium is unique or will be found with all gelling substances 2.

The investigators have completed a study using a modified methylcellulose which was shown to be non-inferior to psyllium.

Our previous studies point to the importance of habitual FODMAP intake which is likely to alter the microbiota, selecting those that can efficiently utilise fructans. The investigators want to understand whether chronic feeding of inulin along with methylcellulose, a gel-forming dietary fibre which persists in the colon, will significantly alter the tolerance to inulin relative to chronic feeding of inulin with a suitable placebo maltodextrin. Maltodextrin is rapidly absorbed in the small bowel and therefore has no effect on colonic fermentation. The investigators plan to run a chronic feeding study in IBS patients and wish to ascertain tolerability of repeated use as previous studies have only provided single doses.

With this in mind, the investigators plan to provide inulin and methylcellulose for daily consumption by healthy adults for a period of two weeks. The intervention will be divided into 3 portions to be taken before breakfast, lunch and supper. In week 1, the portions will contain 2.5 g of both inulin and methylcellulose in 62.5 mL water. In week 2, the portions will contain 5.0 g of both inulin and methylcellulose in 125 mL water. The participants will also follow the same chronic feeding schedule but with a maltodextrin placebo as opposed to methylcellulose, with randomisation of study schedule taking place at screening.

The investigators will use MRI at baseline and at 2 weeks to assess changes in colonic volume and transit utilising high MRI contrast capsules54. The investigators will collect stool samples at baseline and after 1 and 2 weeks of chronic feeding for each study intervention to monitor the expected changes in microbiota. The primary objective is to assess the fermentation of inulin given as a single 15g with or without methylcellulose from the breath hydrogen response at baseline and after the 2 weeks feeding. .

ELIGIBILITY:
Inclusion Criteria:

* • Aged between 18 and 65 years old.

  * Able to give informed consent.
  * Scoring ≤5 (i.e., mild, or less) for symptoms of flatulence, bloating, abdominal pain, loose stool, and hard stool in previous 2 weeks using a modified Gastrointestinal Symptom Rating Scale (5).
  * Agrees to consume the meals provided.
  * Agrees to not smoke during the breath hydrogen sampling period.

Exclusion Criteria:

* • Pregnancy, lactating, or planning pregnancy during the course of the investigation declared by candidate.

  * History declared by the candidate of pre-existing gastrointestinal disorder that may affect bowel function.
  * Reported history of previous resection of the oesophagus, stomach, or intestine (excluding appendix).
  * Intestinal stoma.
  * Any medical condition making participation potentially compromising participation in the study e.g., diabetes mellitus, respiratory disease limiting ability to use breath hydrogen analyser, known intolerance to one of the test substances.
  * Has a body mass index (BMI) value less than 18.5 or greater than 35.
  * Will not agree to follow dietary and lifestyle restrictions required.
  * Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists for the duration of the study (Selective serotonin reuptake inhibitors, low dose tricyclic antidepressants, antihistamines, and oral contraceptive pill will be recorded in the CRF but will not be an exclusion criteria).
  * Participants who are taking antibiotics or probiotics as it might alters gut microbiota.
  * Poor understanding of English language.
  * Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 6.00 AM.
  * Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g., cognitive dysfunction, chaotic lifestyle related to substance abuse.
  * Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Breath hydrogen 0-6 hours post ingestion | 0-6 hours
  Area under curve (AUC) from time 0-6 hours (AUC 0-6) of breath hydrogen (ppm.hour) after consumption of inulin intake.

SECONDARY OUTCOMES:
Symptoms | 14 days
  1) Self-reported symptom scores relating to gastrointestinal tolerance during 2-week chronic feeding period
Breath hydrogen | 0-24 hours
  2) Area under curve (AUC) of breath hydrogen and methane for period 0 - 24hr.
Orocaecal transit | 0- 6 hours
  Time for breath hydrogen to rise > 10ppm over baseline
Whole gut transit time | 0-7 days
  assessed by marker transit
Fecal microbiota | 1 and 2 weeks post dosing
  16s DNA analysis

CONTACTS AND LOCATIONS:
Overall Officials: Robin C Spiller, MD, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Nottingham Digestive Disease Centre, Nottingham, Nottinghamshire
  - Nottingham Digestive Diseases Centre, Nottingham, Please Choose...

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gunn D, Abbas Z, Harris HC, Major G, Hoad C, Gowland P, Marciani L, Gill SK, Warren FJ, Rossi M, Remes-Troche JM, Whelan K, Spiller RC. Psyllium reduces inulin-induced colonic gas production in IBS: MRI and in vitro fermentation studies. Gut. 2022 May;71(5):919-927. doi: 10.1136/gutjnl-2021-324784. Epub 2021 Aug 5. PMID 34353864